CLINICAL TRIAL: NCT05788666
Title: Use of GeriKit to Better Phenotype Older Adults With Ischemic Heart Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 22-00841
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Heart Disease
Keywords: GeriKit; Comprehensive Geriatric Assessment (CGA)
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Geriatric Assessments using GeriKit App (Experimental): Participants will receive comprehensive geriatric assessment via GeriKit app at baseline. All participants will complete a follow-up assessment via phone at 6 months. 20 of the 150 enrolled participants will continue onto a qualitative questionnaire after the completion of the 6-month follow up call.
  Interventions: Procedure: GeriKit Mobile Application

INTERVENTIONS:
Procedure: GeriKit Mobile Application — Digital health app used for comprehensive geriatric assessment (CGA). The app includes a series of brief, well-validated instruments: the MiniCog, 30-Second Chair Stand, Activities of Daily Living, Instrumental Activities of Daily Living, Patient Health Questionnaire (PHQ-9), Mini Nutrition Assessment, 2-Item Fall Screen, and Polypharmacy screen.

SUMMARY:
This study seeks to expand the use of the NYU GeriKit mobile application ("app") in a diverse range of settings to better phenotype older patients, which will enhance both research and patient care.

DETAILED DESCRIPTION:
This is a single-center proof of concept study of geriatric impairments and feasibility metrics through the use of the GeriKit software application in older adults with ischemic heart disease at the NYU Langone Medical Center. The GeriKit mobile application was developed to make geriatric assessment instruments easily accessible to clinicians who do not have subspecialty training in geriatrics. The GeriKit app has been used clinically but is untested in research settings.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 75
2. Currently hospitalized for acute mycardial infarction (AMI), percutaneous coronary intervention (PCI), or coronary artery bypass grafting (CABG); or hospitalized for AMI, PCI, or CABG within the prior 4 weeks
3. Capable of self-consent
4. Understand and are able to perform study procedures in English

Exclusion Criteria:

1. Non-ambulatory
2. Moderate or severe cognitive impairment (operationalized as known diagnosis of dementia)
3. Unable or unwilling to consent
4. Incarcerated
5. Unable to use complete assessments in English
6. Unable to complete geriatric assessment for other reasons

Ages: 75 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Mortality or Hospital Readmission | Month 6
  Binary outcome; determined by review of patient electronic health record (EHR) data at Month 6.

SECONDARY OUTCOMES:
12-Item Short Form Survey (SF-12) Score | Baseline
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality-of-life measure. SF-12 consists of 12 questions that are scored in various ways. The total score range is 12-48; the higher the score, the higher the score, the better the physical and mental health functioning.
12-Item Short Form Survey (SF-12) Score | Month 6
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality-of-life measure. SF-12 consists of 12 questions that are scored in various ways. The total score range is 12-48; the higher the score, the higher the score, the better the physical and mental health functioning.
Seattle Angina Questionnaire Short-Form (SAQ-7) | Baseline
  7-item questionnaire assessing functional status, angina and disease-specific health-related quality of life (HRQoL) over a four-week recall period. Responses generate a summary score ranging from 0-100, where 100 = full health, and 0 = worst health.
Seattle Angina Questionnaire Short-Form (SAQ-7) | Month 6
  7-item questionnaire assessing functional status, angina and disease-specific health-related quality of life (HRQoL) over a four-week recall period. Responses generate a summary score ranging from 0-100, where 100 = full health, and 0 = worst health.

CONTACTS AND LOCATIONS:
Overall Officials: John A. Dodson, MD, MPH, FACC, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: cdhlab@nyumc.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to cdhlab@nyumc.org. To gain access, data requestors will need to sign a data access agreement.